CLINICAL TRIAL: NCT07040930
Title: A Phase Ib Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Subcutaneous Injections of GenSci120 in Healthy Adult Participants in China
Brief Title: Assessment of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Subcutaneous Injections of GenSci120 in Healthy Adult Participants in China.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GenSci120-103
Record Dates: First submitted 2025-06-10; First posted 2025-06-27 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-06

CONDITIONS: Rheumatoid Arthritis
Keywords: phase Ib; healthy adult; multiple subcutaneous injections; GenSci120
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GenSci120 (Experimental): Multiple ascending doses of GenSci120 administered subcutaneously (SC).
  Interventions: Drug: GenSci120
- Placebo (Experimental): Multiple ascending doses of placebo administered subcutaneously (SC).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GenSci120 — a total of 3 doses of the investigational medicinal product (IMP) SC every four weeks (Q4W) at the planned dose level
  Arms: GenSci120
Drug: Placebo — a total of 3 doses of the investigational medicinal product (IMP) SC every four weeks (Q4W) at the planned dose level
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety, tolerability, PK and PD of multiple subcutaneous injections of GenSci120 in a randomized, double-blind, placebo-controlled, multiple-ascending-dose phase Ib trial involving healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-55; ≥3 per gender for each cohort.
2. BMI: 18-30; Weight: ≥50 kg (male), ≥45 kg (female).
3. No clinically significant abnormalities in medical history, physical exam, vital signs, or lab/ECG/pulmonary imaging.
4. Men/WOCBP must use effective contraception throughout study; no plans to conceive; WOCBP must have negative pregnancy test and not breastfeeding. Women of non-childbearing potential: post-hysterectomy/salpingectomy or postmenopausal (FSH >40 IU/L).
5. Able to provide informed consent; willing to comply with all study requirements

Exclusion Criteria:

1. Allergy to GenSci120 or severe allergies.
2. Injection site issues affecting evaluation.
3. Significant medical conditions impacting study outcome.
4. History of malignant tumors, including listed cancers.
5. Seizure history, head injury causing unconsciousness.
6. Psychiatric disorders impairing daily activities or cognitive issues.
7. Severe immunodeficiency (e.g., HIV).
8. Recent trauma, surgery, or GI issues affecting absorption.
9. Recent severe infections or antimicrobial treatments.
10. Live vaccines within a month prior to screening.
11. Abnormal vital signs/ECG: BP extremes, QTcF >450ms.
12. Positive for hepatitis B/C, HIV, syphilis during screening.
13. Positive TB test via IGRA.
14. Recent use of immunosuppressive or targeted therapies.
15. Medication use within 14 days prior to randomization.
16. Participation in other clinical trials recently/currently.
17. Excessive alcohol consumption (over six months).
18. Heavy smoking, unwillingness to quit, positive nicotine tests.
19. Positive drug screen for specific substances.
20. Recent soft/hard drug use within specified periods.
21. Blood donation/product receipt recently or poor venous access.
22. Study staff involved in the trial.
23. Other conditions deemed unsuitable by investigators.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-07-05 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
TEAEs | 169 days
  Incidence and severity of treatment-emergent adverse events
SAEs | 169 days
  Incidence and severity of serious adverse events
CSfadf | 169 days
  Clinically significant changes from baseline

SECONDARY OUTCOMES:
plasma | 169 days
  Concentration of GenSci120 in plasma samples.
AUC0-t, AUC0-∞ | 169 days
  Area under drug concentration-time curve
Tmax | 169 days
  time to maximum concentration
Cmax | 169 days
  maximum concentration
t1/2 | half-life
  169 days
CL/F | apparent clearance
  169 days
V/F | 169 days
  apparent volume of distribution
RO of T cell subset | 169 days
  Receptor occupancy (RO) of T cell subset detected by flow cytometry
cell counts of T cell subset | 169 days
  cell counts of T cell subset detected by flow cytometry
Incidence of ADA | 169 days
  Incidence of anti-drug antibody (ADA) positive positive (if applicable) after GenSci120 administration
Time of ADA | 169 days
  Time of anti-drug antibody (ADA) positive positive (if applicable) after GenSci120 administration

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, M.D., Principal Investigator — Huashan Hospital; Xiaojie Wu, M.D., Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China